CLINICAL TRIAL: NCT00598728
Title: A Global Assessment of Medical Morbidities and Quality of Life Among Survivors of Hodgkin Lymphoma
Brief Title: Quality of Life Among Survivors of Hodgkin Lymphoma
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 05-041
Record Dates: First submitted 2008-01-10; First posted 2008-01-22 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Hodgkin's Disease
Keywords: Survivors; Quality of Life
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- 1: Hodgkin lymphoma Survivors
  Interventions: Behavioral: Quality of Life Questionaires

INTERVENTIONS:
Behavioral: Quality of Life Questionaires — A patient questionnaire, which includes questions on medical morbidities and QOL, will be mailed to participants.

SUMMARY:
The purpose of this study is to collect information on the long-term side effects of treatment for Hodgkin Lymphoma. We hope to study about 500-800 survivors of Hodgkin Lymphoma. We plan to use the findings from this study to better understand Hodgkin Lymphoma survivors' health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven HL Participation in IRB-approved protocols for the first-line treatment of HL between 1975-2000 (IRB #75-104, #75-103, #79-17, #81-103, #90-44, #91-69).
* English speaking

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be recruited from over 800 patients who were enrolled on IRB approved protocols for the firstline treatment of HL between 1975-2000.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2005-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the prevalence of late medical complications among HL survivors | conclusion of study

SECONDARY OUTCOMES:
To study the effect of HL and its treatment on QOL among HL survivors. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: David Straus, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org